CLINICAL TRIAL: NCT04308980
Title: Development and Evaluation of the Effectiveness of Complex Therapy of Steatohepatitis of Various Aetiologies Based on Metabolomic Analysis With the Use of Innovative Medical Nutrition Products
Brief Title: Safety and Tolerability of Novel Medical Nutrition Products for NAFLD Treatment
Acronym: 052920190055
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Russian Academy of Medical Sciences (Other)
Collaborators: Federal State Budgetary Scientific Institution "Federal Research Centre of Nutrition, Biotechnology (Other)
Responsible Party: Principal Investigator, Vasily Isakov, Professor, Russian Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: АААА-А19-119032590090-7/6
Record Dates: First submitted 2020-03-12; First posted 2020-03-16 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: NAFLD; NASH - Nonalcoholic Steatohepatitis
Keywords: diet; nutrition; specialized food product; medical nutrition products; NAFLD; NASH; steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active treatment (Experimental): Patients with verified non-alcoholic fatty liver disease, who signed informed consent to participate in the study and are randomly selected to use specialized medical nutrition product together with diet based on the measured individual requirements in energy and protein intake.
  Interventions: Dietary Supplement: Specialized product for medical nutrition (SPP-1); Behavioral: individualized diet
- Control group (Placebo Comparator): Patients with verified non-alcoholic fatty liver disease, who signed informed consent to participate in the study and are randomly selected to use masked placebo together with diet based on the measured individual requirements in energy and protein intake.
  Interventions: Behavioral: individualized diet

INTERVENTIONS:
Dietary Supplement: Specialized product for medical nutrition (SPP-1) — Patients randomly allocated to this group will use specialized product for medical nutrition (SPP-1). This product contains: soy protein, whey protein concentrate, microcapsulated rapeseed oil, maltodextrin, inulin, Polydextrose, soy lecithin, potassium citrate, magnesium lactate, ω-3 PUFA (docosahexaenoic acid), sweetener mixture (stevia extract, erythritol), natural flavor "Yogurt-vanilla", calcium carbonate, betaine hydrochloride, natural flavor "raspberry", vitamin premix (vitamins a, e, C, D3, B1, B2, B6, B12, PP, folic acid, Pantothenic acid, K1, Biotin), beet juice concentrate, carrageenan, mineral premix (iron, zinc, copper, manganese, iodine, selenium, molybdenum, chromium), alpha-lipoic acid. The product is packed in approved by sanitary rules bags by 30 g. The instant drink obtained by the mixture of the bag content with warm (30-60C) water should be used immediately after being prepared. The daily dose is 1 pack TID
  Arms: Active treatment
Behavioral: individualized diet — All the patients enrolled to the study will be provided with recommendations on diet. Individualized requirements will be calculated based on the results of indirect calorimetry (resting energy expenditures) and measurements of urea in daily urine

SUMMARY:
To the moment, only limited data are present on the efficacy of changes in diet composition of patients with non-alcoholic fatty liver disease (NAFLD). The national database search in the federal registry of specialized products revealed no registered products for medical nutrition for patients with NAFLD. We developed the composition of specialized food products, produced their experimental batches, and performed laboratory studies of their safety, including tests on toxicology and microbiology (which revealed no concerns). Organoleptic studies of the products showed acceptable results. The aim of the present study is to assess safety and tolerability of newly developed specialized products for medical nutrition of patients with non-alcoholic fatty liver diseases in a prospective randomized placebo-controlled trial.

DETAILED DESCRIPTION:
Development of specialized medical products is actual due to the high prevalence of non-alcoholic fatty liver disease (NAFLD), which accounts for 20-30% of the world's population, while non-alcoholic steatohepatitis (NASH) accounts for about 20% of all cases of NAFLD and affects all age groups, including children. Currently, there are no generally accepted and efficient methods to treat the disease. Recommended measures include changes in lifestyle, i.e., weight loss and dietary modifications together with increased physical activity. Pragmatic approaches combining dietary restriction and a progressive increase in aerobic exercise / resistance training are preferable and should be individually tailored. Only general principles of diet modification are strongly recommended, though the evidence of their efficacy is far from excellent. According to EASL 2016 guidelines on NAFLD, there is a need for energy restriction, exclusion of NAFLD-promoting components (processed food, and food and beverages high in added fructose; the macronutrient composition should be adjusted according to the Mediterranean diet) and avoidance of excessive alcohol intake. Only limited data are available on the change of diet composition, including the intake of products with low glycaemic index, containing larger amounts of components with known antioxidant capacity (including vitamins and minerals) and dietary fibre. Still, the use of mentioned components is promising in the regard of their potential to trigger metabolic changes, decrease insulin resistance, inflammatory processes in the liver tissue and excessive lipid accumulation in the liver in patients with NAFLD. The database search in the federal registry of specialized products revealed no specialized products for medical nutrition for patients with NAFLD. Despite some similarities in the pathogenesis of the diseases, specialized medical products for patients with diabetes mellitus are not optimal for patients with fatty liver disease. Based on the published data, medical and biological requirements for specialized product of medical nutrition were formulated. According to them, at an earlier stage of the present work we developed the composition of specialized food products, produced their experimental batches, and performed laboratory studies of their safety, including tests on toxicology and microbiology (which revealed no concerns). Organoleptic studies of the products showed acceptable results. The aim of the present study is to assess safety and tolerability of newly developed specialized products for medical nutrition of patients with non-alcoholic fatty liver diseases in a prospective randomized placebo-controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged from 18 to 75 years inclusive;
* Willingness to participate based on the written informed consent form;
* Documented evidence of non-alcoholic fatty liver disease presence, defined based on the following: steatohepatitis evaluated by liver biopsy taken within 12 months prior to enrolment (when liver biopsy is available, at least a score of 1 in each component of the NAS (steatosis scored 0-3, ballooning degeneration scored 0-2, and lobular inflammation scored 0-3), NAS ≥4, fibrosis stage of 1 or greater and below 4, according to the NASH CRN fibrosis staging system should be present); or ultrasound markers of fatty liver in combination with persistent elevated alanine aminotransferase (ALT; absence of normal value of ALT within the past year), obesity defined by a body mass index (BMI) ≥30, metabolic syndrome (NCEP ATP III definition), type 2 diabetes, or homeostasis model assessment of insulin resistance (HOMA-IR) >6;
* Patients in whom it is safe and practical to proceed with specialized medical food product treatment;
* If a patient is treated with 1 of the following drugs: vitamin E (>400 IU/day), polyunsaturated fatty acids (>2 g/day), or ursodeoxycholic acid; a stable dose from at least 6 months prior to the enrolment;
* For patients with type 2 diabetes, glycaemia must be controlled. If glycaemia is controlled by antidiabetic drugs, change in anti-diabetic therapy must follow these requirements:

  * no qualitative change 6 months prior to randomization (i.e., implementation of a new anti-diabetic therapy) for patients treated with metformin, gliptins, sulfonylureas, sodium/glucose cotransporter (SGLT) 2 inhibitors, glucagon-like peptide (GLP)-1 agonists, or insulin. Dose changes of these medications are allowed in the 6 months prior to randomization, except for GLP-1 agonists, which must remain on stable dose in the 12 months prior to enrolment.
  * no implementation of any antidiabetic drugs before the end of the treatment (day 14).

Exclusion Criteria:

* Pregnant or breast feeding females;
* Liver cirrhosis based on liver histology or liver stiffness measurements (> or equal to 14 kPa), or APRI >or equal to 1; or BARD score > or equal to 2.
* Known chronic heart failure (Grade I to IV of New York Heart Association classification).
* History of efficient bariatric surgery within 5 years prior to enrollment.
* Uncontrolled hypertension during the Screening Period despite optimal antihypertensive therapy.
* Type 1 diabetes patients.
* Patients with haemoglobin A1c [HbA1c] >9.0%.
* Patients with a history of clinically significant acute cardiac event within 6 months prior to Screening
* Weight loss of more than 5% within 6 months prior to Randomization.
* Current or recent history (<5 years) of significant alcohol consumption. For men, significant consumption is defined as higher than 30 g pure alcohol per day. For women, it is typically defined as higher than 20 g pure alcohol per day
* Other well documented causes of chronic liver disease according to standard diagnostic procedures including, but not limited to:

  * positive hepatitis B surface antigen
  * positive hepatitis C Virus (HCV) RNA (tested for in case of known cured HCV infection or positive HCV Ab at Screening)
  * suspicion of drug-induced liver disease
  * alcoholic liver disease
  * autoimmune hepatitis
  * Wilson's disease
  * primary biliary cirrhosis, primary sclerosing cholangitis
  * genetic homozygous haemochromatosis
  * known or suspected hepatocellular carcinoma (HCC)
  * history or planned liver transplant, or current MELD score >12
* Known hypersensitivity to the investigation product or any of its components.
* Patients who are currently participating in, plan to participate in, or have participated in an investigational drug trial or medical device trial containing active substance within 30 days or five half-lives, whichever is longer, prior to Screening.
* Use of the following concomitant medications:

  * Fibrates are not permitted from 2 months before Randomization. Patients that used statins, ezetimibe, or other nonfibrate lipid lowering drugs before Screening may participate if the dosage has been kept constant for at least 2 months prior to Screening.
  * Currently taking drugs that can induce steatosis/steatohepatitis including, but not restricted to: corticosteroids (parenteral & oral chronic administration only), amiodarone (Cordarone), tamoxifen (Nolvadex), and methotrexate (Rheumatrex, Trexall), which are not permitted 30 days prior to Screening and up to end of treatment.
  * Currently taking any medication that could interfere with study medication absorption, distribution, metabolism, or excretion or could lead to induction or inhibition of microsomal enzymes, e.g., indomethacin, which are not permitted from Randomization until end of treatment.
* Patients who have the following associated illnesses or conditions:

  * Any medical conditions that may diminish life expectancy to less than 2 years including known cancers;
  * Evidence of any other unstable or, untreated clinically significant immunological, endocrine, hematological, gastrointestinal, neurological, neoplastic, or psychiatric disease;
  * Mental instability or incompetence, such that the validity of informed consent or ability to be compliant with the study is uncertain.
* patients should not present any of the following biological exclusion criteria:

  * Positive anti-human immunodeficiency virus antibody.
  * Aspartate aminotransferase (AST) and/or ALT >10 x upper limit of normal (ULN).
  * Conjugated bilirubin > 26 umol/l due to altered hepatic function (Gilbert Disease patients are allowed into the study.
  * International normalized ratio >1.40 due to altered hepatic function.
  * Platelet count <100,000/mm^3 due to portal hypertension.
  * Significant renal disease, including nephritic syndrome, chronic kidney disease (defined as patients with markers of kidney damage or estimated glomerular filtration rate [eGFR] of less than 60 ml/min/1.73 m^2).
* Patients for whom participation in the trial is not reasonable according to the opinion of Investigator or in cases when participation in the trial may put the patient at any kind of risk.

The data of patients with evidence or suspected compliance to the provided treatment lower than 80% will be excluded from the analysis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2020-03-20 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Weight change | 14 days
  Assessment of weight before the start of treatment and on the 14th day of treatment. Change will be calculated as a difference from the subtraction of the second measurement from the first.
Change of satiety level | 14 days
  Assessment of satiety will be performed before the start of treatment and on the 14th day of treatment. Change will be calculated as a difference from the subtraction of the second measurement from the first.
Change of hunger level | 14 days
  Assessment of hunger will be performed with the use of the hunger scale before the start of treatment and on the 14th day of treatment. Change will be calculated as a difference from the subtraction of the second measurement from the first.
Presence of adverse events | 14 days
  Assessment of adverse events will be performed before the start of treatment and along the period of treatment.
Change of proportion of fat in body composition | 14 days
  Percent of fat in body composition will be assessed with bioelectrical impedance analysis (bioimpedance, BIA). The change will be calculated as a difference from the subtraction of the second measurement from the first.
Change of proportion of water in body composition | 14 days
  Percent of water in body composition will be assessed with BIA. The change will be calculated as a difference from the subtraction of the second measurement from the first.
Change of lean body weight | 14 days
  Lean weight in body composition will be assessed with BIA. The change will be calculated as a difference from the subtraction of the second measurement from the first.
Change in blood docosahexaenoic acid concentration | 14 days
  High performance liquid chromatography with mass spectrometry analysis of blood samples will be performed to evaluate docosahexaenoic acid concentration before the start of medical food product intake and on the last (14th) day of treatment. The change will be calculated as a difference from the subtraction of the second measurement from the first.
Change in blood hydroxyeycosatetraenoic acid concentration | 14 days
  High performance liquid chromatography with mass spectrometry analysis of blood samples will be performed to evaluate hydroxyeycosatetraenoic acid concentration before the start of medical food product/placebo intake and on the last (14th) day of treatment. The change will be calculated as a difference from the subtraction of the second measurement from the first.

SECONDARY OUTCOMES:
Change of serum glucose concentration | 14 days
  Blood chemistry will be performed before the start of medical food product/placebo intake and on the last (14th) day of treatment. The change will be calculated as a difference from the subtraction of the second measurement from the first.
Change of serum insulin concentration | 14 days
  Blood chemistry will be performed before the start of medical food product/placebo intake and on the last (14th) day of treatment. The change will be calculated as a difference from the subtraction of the second measurement from the first.
Change of serum triglycerides concentration | 14 days
  Blood chemistry will be performed before the start of medical food product/placebo intake and on the last (14th) day of treatment. The change will be calculated as a difference from the subtraction of the second measurement from the first.
Change of serum high-density lipoprotein concentration | 14 days
  Blood chemistry will be performed before the start of medical food product/placebo intake and on the last (14th) day of treatment. The change will be calculated as a difference from the subtraction of the second measurement from the first.
Change of serum low-density lipoprotein concentration | 14 days
  Blood chemistry will be performed before the start of medical food product/placebo intake and on the last (14th) day of treatment. The change will be calculated as a difference from the subtraction of the second measurement from the first.
Change of serum cholesterol concentration | 14 days
  Blood chemistry will be performed before the start of medical food product/placebo intake and on the last (14th) day of treatment. The change will be calculated as a difference from the subtraction of the second measurement from the first.
Change of serum gamma-glutamine transpeptidase (GGT) activity level | 14 days
  Blood chemistry will be performed before the start of medical food product/placebo intake and on the last (14th) day of treatment. The change will be calculated as a difference from the subtraction of the second measurement from the first.
Change of serum alanine amino-transferase (AST) activity level | 14 days
  Blood chemistry will be performed before the start of medical food product/placebo intake and on the last (14th) day of treatment. The change will be calculated as a difference from the subtraction of the second measurement from the first.
Change of serum alanine amino-transferase (ALT) activity | 14 days
  Blood (serum) ALT level will be measured before the start of the product/placebo intake and on the last (14th) day of treatment by blood chemistry. The change will be calculated as a difference from the subtraction of the second measurement from the first.

OTHER OUTCOMES:
Change in concentration of volatile compounds in stool samples | 14 days
  Gas chromatography with mass spectrometry analysis of stool samples obtained before the start of medical food product/placebo intake and on the 14th day of treatment will be performed to evaluate the presence of change in their concentration due to treatment

CONTACTS AND LOCATIONS:
Overall Officials: Vasily Isakov, Professor, Study Chair — FRC Nutrition and Biotechnology
Locations (1):
- Gastroenterology and Hepatology, FRC Nutrition and Biotechnology, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Yes
Blinded IPD data may be available upon request after the study is complete
Supporting Information: Study Protocol, ICF, CSR
Time Frame: After study completion within 2 years
Access Criteria: Upon request
URL: http://ion.ru

REFERENCES:
- [Background] European Association for the Study of the Liver (EASL); European Association for the Study of Diabetes (EASD); European Association for the Study of Obesity (EASO). EASL-EASD-EASO Clinical Practice Guidelines for the management of non-alcoholic fatty liver disease. J Hepatol. 2016 Jun;64(6):1388-402. doi: 10.1016/j.jhep.2015.11.004. Epub 2016 Apr 7. No abstract available. PMID 27062661
- [Background] Vernon G, Baranova A, Younossi ZM. Systematic review: the epidemiology and natural history of non-alcoholic fatty liver disease and non-alcoholic steatohepatitis in adults. Aliment Pharmacol Ther. 2011 Aug;34(3):274-85. doi: 10.1111/j.1365-2036.2011.04724.x. Epub 2011 May 30. PMID 21623852
- [Background] Barrera F, George J. The role of diet and nutritional intervention for the management of patients with NAFLD. Clin Liver Dis. 2014 Feb;18(1):91-112. doi: 10.1016/j.cld.2013.09.009. Epub 2013 Oct 24. PMID 24274867
- [Background] Zelber-Sagi S, Ratziu V, Oren R. Nutrition and physical activity in NAFLD: an overview of the epidemiological evidence. World J Gastroenterol. 2011 Aug 7;17(29):3377-89. doi: 10.3748/wjg.v17.i29.3377. PMID 21876630
- [Background] Arab JP, Candia R, Zapata R, Munoz C, Arancibia JP, Poniachik J, Soza A, Fuster F, Brahm J, Sanhueza E, Contreras J, Cuellar MC, Arrese M, Riquelme A. Management of nonalcoholic fatty liver disease: an evidence-based clinical practice review. World J Gastroenterol. 2014 Sep 14;20(34):12182-201. doi: 10.3748/wjg.v20.i34.12182. PMID 25232252
- [Background] Boden G. High- or low-carbohydrate diets: which is better for weight loss, insulin resistance, and fatty livers? Gastroenterology. 2009 May;136(5):1490-2. doi: 10.1053/j.gastro.2009.03.019. Epub 2009 Mar 21. No abstract available. PMID 19318102
- [Background] Argo CK, Patrie JT, Lackner C, Henry TD, de Lange EE, Weltman AL, Shah NL, Al-Osaimi AM, Pramoonjago P, Jayakumar S, Binder LP, Simmons-Egolf WD, Burks SG, Bao Y, Taylor AG, Rodriguez J, Caldwell SH. Effects of n-3 fish oil on metabolic and histological parameters in NASH: a double-blind, randomized, placebo-controlled trial. J Hepatol. 2015 Jan;62(1):190-7. doi: 10.1016/j.jhep.2014.08.036. Epub 2014 Sep 6. PMID 25195547
- [Background] Ryan MC, Itsiopoulos C, Thodis T, Ward G, Trost N, Hofferberth S, O'Dea K, Desmond PV, Johnson NA, Wilson AM. The Mediterranean diet improves hepatic steatosis and insulin sensitivity in individuals with non-alcoholic fatty liver disease. J Hepatol. 2013 Jul;59(1):138-43. doi: 10.1016/j.jhep.2013.02.012. Epub 2013 Feb 26. PMID 23485520
- [Derived] Sasunova AN, Morozov SV, Sobolev RV, Isakov VA, Kochetkova AA, Vorobyeva IS. [Efficacy of newly developed food for special dietary use in the diet of patients with non-alcoholic steatohepatitis]. Vopr Pitan. 2022;91(2):31-42. doi: 10.33029/0042-8833-2022-91-2-31-42. Epub 2022 Mar 14. Russian. PMID 35596633
- See also: Information about institution where the study is performed — http://ion.ru